CLINICAL TRIAL: NCT06365749
Title: Exome Sequencing Explored the Genetic Characteristics Congenital Hearing Loss in Chinese Population
Brief Title: Genetic Feature of Congenital Hearing Loss in Chinese Population
Status: Not yet recruiting | Type: Observational
Sponsor: Dan Bing (Other)
Responsible Party: Sponsor-Investigator, Dan Bing, associate professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20221228
Record Dates: First submitted 2023-11-21; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Congenital Hearing Loss; Congenital Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample with DNA will be collected from heel prick or cord blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonate with hearing loss: Neonates who failed in the neonatal hearing screening programs, including oto-acoustic emissions and automated auditory brain stem response.

SUMMARY:
Congenital hearing loss, as well as hearing loss present at birth, is one of the most common chronic conditions in children, with a prevalence of permanent bilateral hearing loss of 2.83 per 1000 children of primary school age, which is mainly caused by genetic factors. The goal of this observational study is to learn about novel causative genes in infants with hearing loss in the Chinese population. The main problem it aims to deal with are:

* to present the genetic characteristics of the infant with hearing loss in the Chinese population
* to build up a prognostic model base on diverse data.

Participants will be asked to receive audiological tests and collection of the peripheral blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Age up to 6 months
* Fail in the neonatal hearing screening programs, including oto-acoustic emissions and automated auditory brain stem response
* Promise to complete the tests required at baseline and follow-ups by the legal representative
* Informed consent by the legal representative

Exclusion Criteria:

* Congenital infections related to acquired or congenital hearing loss, including rubella virus, cytomegalovirus, herpes simplex virus, rubella virus, toxoplasma gondii and treponema pallidum infections
* Other explicit otologic conditions which could induce hearing loss, including cerumen, otitis media, congenital middle ear abnormalities, microtia and external ear abnormalities
* A drug with ototoxicity usage during pregnancy
* Other severe congenital anomalies

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates who were offered neonatal hearing screening programs at Tongji hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-23 (Estimated); Primary Completion 2026-11-23 (Estimated); Study Completion 2026-11-23 (Estimated)

PRIMARY OUTCOMES:
Whole exome sequencing data | Baseline
  DNA of neonate extracted from blood sample by heel prick or collection of cord blood will be perform whole exome sequencing to present genetic features. By sequencing all protein-coding regions, WES uncovers mutations that can inform diagnostic, therapeutic, and preventive strategies. Key outcome measures from WES include the detection of single nucleotide polymorphisms, insertions, deletions, and structural variants. These outcomes are critical for diagnosing genetic disorders, personalizing treatments, and assessing disease risk. The analysis involves aligning reads to a reference genome, calling variants, and interpreting their clinical significance. WES data thus serves as a cornerstone in genetic research and personalized medicine, enabling a deeper understanding of the genetic underpinnings of diseases and tailoring healthcare approaches to individual genetic profiles.

SECONDARY OUTCOMES:
TEOAE-based otoacoustic emissions test outcome measure | Baseline
  In analyzing Transient Evoked Otoacoustic Emissions (TEOAE), key factors include response reproducibility, which indicates consistent cochlear responses, and signal-to-noise ratio (SNR), where a value above 3 dB suggests clear cochlear emissions against background noise. The Response Spectrum provides a frequency-specific look at cochlear performance, essential for identifying potential hearing issues. A 'Pass' in the TEOAE test denotes normal cochlear function, while a 'Refer' indicates the need for further hearing evaluations.
Auditory brainstem response testing | Baseline
  In auditory brainstem response (ABR) testing, waveform reproducibility and waveform latency, especially of Wave V, are key. High reproducibility indicates reliable signal transmission, suggesting a healthy auditory system. Appropriate latency for Wave V indicates efficient signal processing. Frequency-Specific Responses highlight the brainstem's reaction across different sound frequencies, aiding in identifying potential issues. 'Normal' ABR results reflect functional auditory pathways, while 'Abnormal' ones prompt further investigation.
Acoustic impedance | Baseline
  Acoustic impedance, a critical parameter in sound wave dynamics, quantifies a medium's opposition to sound propagation, expressed as the ratio of acoustic pressure to particle velocity. This parameter is shaped by the medium's density and the speed of sound through it, pivotal for understanding sound behavior in various environments. In audiology, specifically in tympanometry, impedance measurements diagnose middle ear conditions by assessing how sound waves are absorbed or reflected, revealing conditions like effusion or tympanic membrane perforations. The results are typically classified into Jerger types, which categorize middle ear function based on the impedance curve's shape and peak characteristics, providing a detailed insight into middle ear health. High impedance may indicate obstructions or stiffness in the middle ear, while low impedance could suggest perforations or discontinuities.
Audiogram | 4 years follow up
  Pure-tone threshold testing is a cornerstone of audiological assessment, used to determine the softest level at which an individual can hear sounds of specific frequencies. During the test, pure tones of various frequencies are presented through headphones or earphones to one ear at a time, or through a speaker for bone conduction testing. The process begins at an audible level, gradually decreasing until the sound is no longer heard, then slightly increasing until it is heard again. This method helps identify the threshold, or the lowest level at which a sound is perceived 50% of the time for each frequency tested, typically ranging from low (250 Hz) to high (8000 Hz) frequencies.